CLINICAL TRIAL: NCT07113899
Title: HOPE AND ACCEPTANCE AT THE END OF LIFE - IMPACT OF SPIRITUALITY ON PALLIATIVE CARE PATIENTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unidade Local de Saúde de Coimbra, EPE (Other)
Responsible Party: Principal Investigator, Lutenio Junior, Principal Investigator, Unidade Local de Saúde de Coimbra, EPE
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CE-190/2024
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2024-12

CONDITIONS: Hope; Acceptance; Spirituality
Keywords: hope; acceptance; spirituality; end of life; palliative care
MeSH Terms: conditions — Death

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ECSCP (Experimental): Patients visited at home by the community palliative care support team
  Interventions: Other: Approach to spirituality through hope and acceptance
- CSP (No Intervention): Patients with follow-up consultations by primary health care

INTERVENTIONS:
Other: Approach to spirituality through hope and acceptance — This study is a prospective longitudinal research study. The sample consisted of two groups: the Intervention Group, which included patients from the community palliative care support team (ECSCP-BM), and the Control Group, with primary health care selected patients from the family health units Nautilus and Coimbra Centro (CSP), with serious illness, comorbidities, and a poor prognosis. The patients chosen from ECSCP-BM were made up only of new patients referred to the team without any prior home consultations. The first questionnaire application took place during the first visit, and the second one was administered fourteen days later. The Primary Health Care patients were selected by invitation, and the questionnaire was administered. It included sociodemographic data, clinical data, the Herth Hope Index and open questions.
  During the palliative care team's home visit, spirituality was addressed in in the clinical history through the assessment of hope and acceptance.
  Arms: ECSCP

SUMMARY:
This study aims to evaluate the hope and acceptance among patients visited by the Equipa Comunitária de Suporte em Cuidados Paliativos do Baixo Mondego. This study is a prospective longitudinal research study. The sample consisted of two groups: the Intervention Group, which included patients from the network of the Equipa Comunitária de Suporte em Cuidados Paliativos do Baixo Mondego (ECSCP-BM), and the Control Group, with selected patients from Unidade de Saúde Familiar Nautilus e Unidade de Saúde Familiar Coimbra Centro, with serious illness, comorbidities, and a poor prognosis. The patients chosen from ECSCP-BM were made up only of new patients referred to the team without any prior home consultations. The first questionnaire application took place during the first visit, and the second one was administered fourteen days later. The Primary Health Care patients were selected by invitation, and the questionnaire was administered. It included sociodemographic data, clinical data, the Herth Hope Index - PT and open questions.

ELIGIBILITY:
Inclusion Criteria:

* new referrals made by the family doctor to the community palliative care support team (which integrated the patient into the palliative care team network for the first time) - for the intervention group
* patients registered at the Nautilus Family Health Unit or Coimbra Centro Family Health Unit with serious pathology, comorbidities and reserved prognosis - for the control group

Exclusion Criteria:

* age under 18
* pregnancy
* altered state of consciousness or dementia
* low level of education

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Hope | 5 months
  Participants answered questions on the Hope Scale. There were 9 questions with 4 possible answers. Each answer was scored from 1 to 4. The maximum score on the scale was 36.
Acceptance | 5 months
  Participants answered three open-ended questions to assess their acceptance. These questions were asked to the control group and at the first assessment of the intervention group. At the second assessment of the intervention group, after 14 days, a fourth question was also asked, assessing the team's intervention during those 14 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Lutenio Soares Faria Junior, Coimbra, Coimbra District, Portugal